CLINICAL TRIAL: NCT06015516
Title: Randomised, Crossover Bioavailability Clinical Trial of Oral Minoxidil 1 MG, After Single and Multiple Dose Administration to Healthy Volunteers Under Fasting Conditions.
Brief Title: Bioavailability Clinical Trial of Oral Minoxidil 1 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: P23112a; 2023-503796-14-00 (Other: EU CTIS)
Record Dates: First submitted 2023-05-31; First posted 2023-08-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Bioavailability; Clinical trial; minoxidil
MeSH Terms: interventions — Minoxidil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Test: Oral minoxidil 1 mg tablets (Experimental): Participants will be administered one tablet of oral minoxidil 1mg once a day, orally, after fasting for at least 10 hours, with 240 mL or 8 Oz. of water, and fasting for a further 5 hours.
  Interventions: Drug: Minoxidil Tablets
- Treatment Reference: Regaxidil 20 mg/ml (2%) topical solution (Active Comparator): Participants will be administered topically on the scalp after fasting for at least 10 hours pre-dose and 5 hours post-dose. After the administration subject should not wash her head for at least 5 hours. Each one mL dose of 2% topical minoxidil will be carefully measured to provide 20 mg of minoxidil using the syringe provided with each bottle.
  Interventions: Drug: Minoxidil topical solution 20 mg/ml

INTERVENTIONS:
Drug: Minoxidil Tablets — Since oral minoxidil is a new formulation and, according to the recommendations of the Regulatory Authorities, it is considered appropriate to carry out a multiple dose study to evaluate and to compare the bioavailability between both formulations (oral versus topical solution), measuring the plasma concentrations of minoxidil.
  Achievement of steady-state is assessed by comparing at least three pre-dose concentrations for each formulation, as half-life of minoxidil is around 4 hours, we will administered 5 doses in each period.
  Arms: Treatment Test: Oral minoxidil 1 mg tablets
Drug: Minoxidil topical solution 20 mg/ml — Since oral minoxidil is a new formulation and, according to the recommendations of the Regulatory Authorities, it is considered appropriate to carry out a multiple dose study to evaluate and to compare the bioavailability between both formulations (oral versus topical solution), measuring the plasma concentrations of minoxidil.
  Achievement of steady-state is assessed by comparing at least three pre-dose concentrations for each formulation, as half-life of minoxidil is around 4 hours, we will administered 5 doses in each period.
  Arms: Treatment Reference: Regaxidil 20 mg/ml (2%) topical solution

SUMMARY:
The goal of this clinical trial is to learn about the pharmacokinetic profile (behaviour of the drug in the body) of a new oral formulation of minoxidil administered in healthy volunteers.

The main question that is to answer is to evaluate the bioavailability of the oral test formulation of minoxidil. The secondary onjectives is to compare it with the formulation already on the market (i.e . Regaxidil® 20 mg/mL cutaneous solution).

It is planned that 14 healthy female volunteers of legal age (without any known pathology) participate in the study. The expected duration of the study is approximately 23-56 days.

Each volunteer that decide to participate in this study will be sequentially administered one of the formulations planned for the study: either the test formulation (oral minoxidil tablets of 1 mg, developed by Industrial Farmacéutica Cantabria, S.A.), or the reference formulation (minoxidil skin solution, 20 mg/mL, marketed by Industrial Farmacéutica Cantabria, S.A.). After five days of administration of one of the study formulations, at least 7 days will elapse before starting an additional five days of administration of the other study formulation that had not been administered in the first sequence. Assignment to this sequence of administration of the study formulations (oral formulation or topical solution) shall be completely randomised.

In each of these sequential periods of five days of administration of the study formulations, the concentration of minoxidil will be quantified in blood samples, which will be taken from each of the volunteers at certain times after the administration of the medication. These blood analyses will enable to determine the parameters that define the pharmacokinetic profile of the new oral formulation under study.

DETAILED DESCRIPTION:
This is a phase I, oral multiple-dose, open-label, crossover and randomized clinical trial, 2 sequences, 2 periods, in which subjects will be hospitalized from 10 h before to 12 hours after the first and fifth doses under fasting conditions in both periods.

The study will be blinded only for the plasma concentrations determination of minoxidil.

It is planned to include 14 healthy women volunteers, aged from 18 to 55 years old. The overall duration of the study is estimated at 24-56 days, from recruitment of the volunteers to the last examination.

The test drug is minoxidil 1 mg tablets, manufactured by Industrial Farmacéutica Cantabria, S.A. It will be administered a total of five 1 mg doses (once a day) per oral, under fasting conditions. The reference drug is minoxidil 20 mg/ml (2%) topical solution, marketed in Spain by Industrial Farmacéutica Cantabria, S.A., under the name the trade name of Regaxidil®. It will be applied five 1 mL doses (once a day) topical route, under fasting conditions.

Each one of the subjects will receive a daily dose during five days of minoxidil test or reference in each one of the two periods according to the corresponding randomization sequence, after at least 7 days washout period between each one of admission days.

The main objective is to evaluate the relative bioavailability of the oral test formulation of minoxidil 1 mg after single dose and multiple dose (at steady state). The bioavailability of oral formulation will be evaluated from the AUC0-t and Cmax for single dose on the first administration day and AUC(0-τ)SS, Cmax,ss and Cτ,ss on the steady state of minoxidil. Tmax and Tmax,ss and fluctuation of minoxidil will be also calculated. All the pharmacokinetic parameters will be calculated from the plasma concentrations of minoxidil of the formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Women, who after receiving information about the study design, the objectives, the possible risks that could be derived from it and the fact that they can refuse to collaborate at any time, give their written informed consent to participate in the study.
2. Aged from 18 to 55 years old.
3. No clinically significant organic or psychic conditions.
4. No clinically significant abnormalities in medical records and physical examination.
5. No clinically significant abnormalities in haematology, coagulation, biochemistry, serology (Ag HBs, HC antibodies, HIV antibodies) and urinalysis.
6. No clinically significant abnormalities in vital signs and electrocardiogram.
7. Women of child-bearing potential age women participating in the study will compromise to use a high effective contraceptive method or will be abstinent during their participation in the study.

Exclusion Criteria:

1. Subjects affected by an organic or psychic condition. Before a volunteer is included, all the safety parameters defined in points 7.3 will be considered. Those who present clinically significant analytical alterations and in whom biochemical kidney and/or liver damage markers are outside the normal range applied by the laboratory will be excluded [GOT, GPT and/or GGT >2.5*ULN and total bilirrubin >1.5*ULN (total bilirrubin >1.5*ULN is acceptable if the direct bilirrubin is <35%)].
2. Subjects who have received prescribed pharmacological treatment in the last 15 days or abstinent of medication in the 48 hours prior to receiving the study medication, but women are allowed taking contraceptives. Contraceptive methods must be used at least 4 weeks prior to entry visit and not to be changed for the duration of the study.
3. Subjects with body mass index (weight (kg)/height2 (m2)) outside the 18.5-30.0 range.
4. History of sensitivity to any drug.
5. Positive drug screening for cannabis, opiates, cocaine and amphetamines.
6. Smoker.
7. Daily consumers of alcohol and/or acute alcohol poisoning over the last week.
8. Having donated blood in the last month before start of the study.
9. Pregnant or breastfeeding women.
10. Participation in another study with administration of investigational drugs in the previous 3 months (if the study was conducted with drug substances marketed in Spain, a period of at least 1 month or 5 half lives, what is longer, will be considered).
11. Inability to follow the instructions or collaborate during the study.
12. History of difficulty in swallowing
13. Alterations on the scalp such as erythema, dryness or any other condition that at investigator criteria could affect the absortion of the topical solution.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to the last determination (AUC0-t and AUC(0-τ)ss) for minoxidil. | Day 0 (pre-dose) and at multiple time-points (up to day 5) post-dose.
  According to the recommendations of the regulatory authorities, for the analysis of the compared bioavailability of the formulations from single dose and under steady-state conditions, the primary endpoint will be the area under the curve during a dosage interval (AUC0-t and AUC(0-τ)ss) calculated using the linear trapezoidal method, maximum plasma concentration (Cmax and Cmax,ss) and concentration at the end of the dosing interval (Cτ,ss) at steady state calculated from the plasma concentrations of minoxidil.
Maximum observed plasma concentration (Cmax and Cmax,ss) for minoxidil from time zero to the last determination at steady state (Cτ,ss). | Day 0 (pre-dose) and at multiple time-points (up to day 5) post-dose.
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
  According to the recommendations of the regulatory authorities, for the analysis of the compared bioavailability of the formulations from single dose and under steady-state conditions, the primary endpoint will be the area under the curve during a dosage interval (AUC0-t and AUC(0-τ)ss) calculated using the linear trapezoidal method, maximum plasma concentration (Cmax and Cmax,ss) and concentration at the end of the dosing interval (Cτ,ss) at steady state calculated from the plasma concentrations of minoxidil.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) for both minoxidil formulations. | Day 0 (pre-dose) and at multiple time-points (up to day 5) post-dose.
  The relative bioavailability of the oral test formulation of minoxidil is obtained by analysing the AUC from plasma concentrations of both formulations of minoxidil (oral and topical solution) and then these will compared.
Maximum Plasma Concentration (Cmax) and Peak Cmax steady state for both minoxidil formulations. | Day 0 (pre-dose) and at multiple time-points (up to day 5) post-dose.
  The relative bioavailability of the oral test formulation of minoxidil is obtained by analysing the fhe peak concentration (Cmax and Cmax,ss) from plasma concentrations of both formulations of minoxidil (oral and topical solution) and then these will compared.
To evaluate the safety and tolerability of oral minoxidil . | Day 0 (pre-dose) and at multiple time-points (up to day 5) post-dose.
  The safety profile of oral minoxidil will be evaluated by analysing the incidence of adverse events of the oral test formulation compared the commercial formulation. The safety parameters will be expressed individually as mean values +/- standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Ochoa Mazarro, Principal Investigator — Clinical Trial Unit, Clinical Pharmacology Department Hospital Universitario de La Princesa (Madrid, Spain)
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messenger AG, Rundegren J. Minoxidil: mechanisms of action on hair growth. Br J Dermatol. 2004 Feb;150(2):186-94. doi: 10.1111/j.1365-2133.2004.05785.x. PMID 14996087
- [Background] Shamsaldeen OS, Al Mubki T, Shapiro J. Topical agents for hair growth promotion: what is out there? Skin Therapy Lett. 2013 Jun;18(4):5-7. PMID 24310642
- [Background] Vano-Galvan S, Pirmez R, Hermosa-Gelbard A, Moreno-Arrones OM, Saceda-Corralo D, Rodrigues-Barata R, Jimenez-Cauhe J, Koh WL, Poa JE, Jerjen R, Trindade de Carvalho L, John JM, Salas-Callo CI, Vincenzi C, Yin L, Lo-Sicco K, Waskiel-Burnat A, Starace M, Zamorano JL, Jaen-Olasolo P, Piraccini BM, Rudnicka L, Shapiro J, Tosti A, Sinclair R, Bhoyrul B. Safety of low-dose oral minoxidil for hair loss: A multicenter study of 1404 patients. J Am Acad Dermatol. 2021 Jun;84(6):1644-1651. doi: 10.1016/j.jaad.2021.02.054. Epub 2021 Feb 24. PMID 33639244
- See also: Summary of Product Characteristics (SmPC): Minoxidil 20 mg/ml solución cutánea — http://cima.aemps.es/cima/dochtml/ft/57597/FT_57597.html
- See also: Summary of Product Characteristics (SmPC): Minoxidil 10 mg tablets. — http://cima.aemps.es/cima/dochtml/ft/55636/FT_55636.html